CLINICAL TRIAL: NCT06541093
Title: Phase 1 Proof-of-Concept Study to Evaluate the Safety and Immunogenicity of a Priming VaccinationRegimen of Uvax Bio's Glycan Trimmed HIV-1 Vaccine (UVAX-1107) With CpG 1018®/Aluminum HydroxideAdjuvant in Healthy Adults (25-55 Years), Followed by Boosting Vaccination Regimen Using UVAX-1107 orWildtype Non-Glycan Trimmed HIV-1 Vaccine (UVAX-1197) With CpG 1018®/Aluminum Hydroxide Adjuvant
Brief Title: Study to Evaluate the Safety and Immunogenicity of an HIV-1 Vaccine Regimen of Adjuvanted UVAX-1107 Followed by Adjuvanted UVAX-1107 or Adjuvanted UVAX-1197 in Healthy Subjects Aged 25-55 Years.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Uvax Bio LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UVAX-HIV-101
Record Dates: First submitted 2024-06-21; First posted 2024-08-07 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: AIDS/HIV - RelatedDisease Associated With AIDS; Vaccine-Preventable Diseases; HIV Infections
Keywords: Vaccine; HIV; AIDS; Prevention
MeSH Terms: conditions — Vaccine-Preventable Diseases; HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- UVAX-1107 half dose + UVAX-1197 half dose boost (Experimental)
  Interventions: Biological: UVAX-1107; Biological: UVAX-1197
- UVAX-1107 full dose + UVAX-1197 full dose boost (Experimental)
  Interventions: Biological: UVAX-1107; Biological: UVAX-1197
- UVAX-1107 full dose + UVAX-1107 full dose boost (Experimental)
  Interventions: Biological: UVAX-1107
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: UVAX-1107 — Novel HIV-1 protein nanoparticles vaccine candidate (WT) mixed with Aluminum Hydroxide (AH) and CpG 1018 adjuvants
  Arms: UVAX-1107 full dose + UVAX-1107 full dose boost; UVAX-1107 full dose + UVAX-1197 full dose boost; UVAX-1107 half dose + UVAX-1197 half dose boost
Biological: UVAX-1197 — Novel HIV-1 protein nanoparticles vaccine candidate (GT) mixed with Aluminum Hydroxide (AH) and CpG 1018 adjuvants
  Arms: UVAX-1107 full dose + UVAX-1197 full dose boost; UVAX-1107 half dose + UVAX-1197 half dose boost
Other: Placebo — Saline injection
  Arms: Placebo

SUMMARY:
This is a first in human testing of novel HIV-1 protein nanoparticles vaccine candidates, UVAX-1107 and UVAX-1197 mixed with Aluminum Hydroxide (AH) and CpG 1018 adjuvants. After meeting all eligibility criteria, approximately 34 participants will receive a 4-dose vaccination regimen of either 2 priming vaccinations of UVAX-1107 followed by 2 boosting vaccinations of UVAX-1197, or 4 doses of UVAX-1107, or placebo. Subject participation is expected to last up to 374 days, including up to a 30-day screening period and a 337-day study period during which subjects will be followed for safety and immunogenicity outcomes.

DETAILED DESCRIPTION:
This is a first in human testing of a novel HIV-1 vaccine candidate. Both UVAX-1197 and UVAX-1107 are protein nanoparticle vaccines displaying an uncleaved, prefusion-optimized (UFO) envelope (Env) glycoprotein from HIV-1 BG505 (BG505-UFO). The UVAX-1197 displays fully glycosylated UFO Env trimers with wildtype glycans (WT). UVAX-1107 is derived from UVAX-1197 by enzymatic "glycan trimming" (GT) of N-linked glycans in order to better expose major neutralizing epitopes on the surface of BG505-UFO Env to immune recognition. The optimized vaccine immunogens will be mixed with Aluminum Hydroxide (AH) and CpG 1018 adjuvants to enhance the immune response. Subject participation is expected to last up to 374 days, including up to a 30-day screening period and a 337-day study period.

Part 1 of the study will be a safety lead-in cohort in which 4 participants will receive 2 priming vaccinations of a half dose of adjuvanted UVAX-1107 (administered in 0.5ml intramuscular injection) on Days 1 and 57 followed by boosting vaccinations of a half dose of adjuvanted UVAX-1197 on Days 141 and 225, administered as intra-muscular (IM) injections. Safety will be reviewed after subjects in Part 1 reach Day 8, prior to opening Part 2.

A separate group of participants will be enrolled in Part 2 of the study. Participants in Part 2 will be randomized to the following treatment arms to receive either:

* Priming vaccinations of adjuvanted UVAX-1107 (full dose, administered in 0.5ml intramuscular injection) on Days 1 and 57 followed by boosting vaccinations of adjuvanted UVAX-1197 (full dose, administered in 0.5ml intramuscular injection) on Days 141 and 225.
* Priming vaccinations of adjuvanted UVAX-1107 (full dose) on Days 1 and 57 followed by boosting vaccinations of adjuvated UVAX-1107 (full dose) on Days 141 and 225.

When Part 2 of the study opens, 5 sentinel participants (2 from each of the active treatment groups and 1 from the placebo group) will be randomized. Safety will be reviewed after these first 5 Part 2 participants reach Day 8 prior to opening randomization to the remaining participants in Part 2.

Vaccinations will be administered by trained staff at the study site(s) according to site's SOPs. Details regarding dosing, including the dose administered, arm, and the date and time of dosing, will be recorded in the subjects source notes and electronic case report form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 25-55 years of age, inclusive, at screening.
2. Stable health status, as established by physical examination and medical history.
3. Capable of providing written informed consent.
4. Female participants of reproductive potential must be non-pregnant and non lactating, and if of child-bearing potential must agree to be heterosexually inactive from at least 21 days prior to enrolment (Day 1)and through 90 days following last study vaccination or agrees to consistently use highly effective method of birth control and refrain from donating oocytes from at least 21 days prior to enrolment and through 90 days following last study vaccination.
5. Male participants must:

   1. Agree not to donate sperm from the time of signing consent until at least 90 days after the last dose of study drug.
   2. If engaging in sexual intercourse with a female partner who could become pregnant, must agree to use adequate contraception until at least 90 days after the last dose of study drug.
   3. If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, must agree to use a condom.

Exclusion Criteria:

1. Chronic illness being treated actively and with evidence of recent adjustments in medications for worsening or fluctuating symptoms in the past 3 months, or hospitalizations / procedural interventions in the past 6 months.
2. Body mass index (BMI) of less than 17 and greater than 32 kg/m2 at screening.
3. Vital signs grading greater than 1 at screening
4. Toxicity grading greater than 1 for screening laboratory test results.
5. Any abnormal, clinically significant ECG result at screening.
6. High risk of contracting HIV.
7. History of cancer (malignancy) in the last 10 years.
8. Use of narcotic/illicit drugs or a history of drug/alcohol abuse within the past 2 years.
9. Has donated blood or suffered from blood loss of more than 450 mL (1 unit of blood) within 60 days prior to screening, or donated plasma within 14 days prior to screening.
10. Receipt of immunoglobulin, blood-derived products, high dose systemic corticosteroids, or other immunosuppressant drugs within 90 days prior to Day 1 or who expect to receive immunoglobulin or another blood product during the study.
11. Receipt of a licensed or emergency/provisional approval vaccine within the last 30 days prior to Day 1.
12. Known hypersensitivity to any component of the study vaccines, including history of anaphylaxis or other significant allergy in the opinion of the Investigator.
13. Any autoimmune or immunodeficiency disease/condition (inherited or iatrogenic) or chronic hematologic disorder (anemia, sickle cell, thalassemia).
14. Evidence of HIV, positive hepatitis B surface antigen or core antibody or hepatitis C antibodies by screening test.
15. Any chronic or degenerative neurological disease or history of significant neurological disorder.
16. Evidence of cardiovascular, pulmonary, renal, hepatobiliary disease or any other baseline condition (history and medication review) that has required active treatment or intervention.
17. Evidence of major depression disorder not well controlled in the past 2 years or history of suicidal ideation or attempt in the past 2 years.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
To assess local and systemic reactogenicity following vaccination (Day 1 to Day 8, inclusive) following each vaccination. | Days 1 through Day 7 after each vaccination.
  Reactogenicity (local and systemic) will be recorded by the subject using a daily diary after vaccination andfor 6 consecutive days thereafter.
To determine if antibody responses are induced at 2 weeks after each vaccination using anti-HIV-1 protein IgG. | Pre-vaccination timepoints (Day 1, Day 57, Day 141 and Day 225) and ~2 weeks after each vaccination (Day15, Day 71, Day 155 and Day 239) and Day 337 post enrolment/End of study (EOS).
  Serum samples will be collected at specified timepoints for HIV-1-specific IgG titers

SECONDARY OUTCOMES:
To assess serious adverse events (SAEs) or adverse events of special interest (AESI) attributed to vaccination. | At all visits, Day 1, Day 8, Day 15, Day 29, Day 57, Day 64, Day 71, Day 85, Day 141, Day 148, Day 156, Day 169,Day 225, Day 232, Day 239, Day 253 and Day 337 post enrolment/End of Study (EOS).
  As the proposed trial (UVAX-HIV-101) will be the first study of UVAX-1197 and -1107 in humans, there is currently no data regarding AEs associated with either UVAX-1197 or -1107 in humans. UVAX-1197 and -1107 have been administered in animals without significant adverse reactions being observed. Based on preclinical experience and AEs generally observed in other intramuscular administered vaccines using a similar development platform, the vaccinations are expected to result in mild to moderate local reactions and/or systemic reactions. These AEs will be assessed via clinical examination at the reference timepoints and via the use of a subject diary for the 7 days following each vaccination.
To describe occurrence of Medically Attended Adverse Events (MAAEs). | On pre- and post-dose Day 1, Day 8, Day 15, Day 29, pre- and post-dose Day 57, Day 64, Day 71, Day 85,pre- and post-dose Day 141, Day 148, Day 156, Day 169, pre- and post-dose Day 225, Day 232, and Day 253
  MAAEs (e.g. any AEs that are evaluated by a healthcare professional either at the site or within the community) will be reported from Day 1 through 28 days after the last vaccination was received. They will be assessed using study-specific questionnaire, clinical examination and data-linkage to medical records. These AEs will be assessed via clinical examination at the reference timepoints and via the use of a subject diary for the 7 days following each vaccination.
To describe occurrence of treatment emergent adverse events (TEAEs) | Endpoint will evaluate TEAEs reported until Day 29 following each vaccination (Day 1, Day 8, Day 15, Day 29,post-dose Day 57, Day 64, Day 71, Day 85, post-dose Day 141, Day 148, Day 156, Day 169, post-dose Day225, Day 232, and Day 253).
  TEAEs (e.g. any AEs that occur after the study product has been administered) will be reported throughout the study period until Day 253 (28 days following the last dose) .They will be assessed, using study-specific questionnaire, clinical examination and data-linkage to medical records. These AEs will be assessed via clinical examination at the reference timepoints and via the use of a subject diary for the 7 days following each vaccination
To describe occurrence of laboratory-related adverse events from pre-vaccination to 7 days following each vaccination. | Screening visit, Day 8, pre-dose Day 57, Day 64, pre-dose Day 141, day 148, pre-dose Day 225, Day 239 and Day 337 post-enrolment/End of Study (EOS)
  Clinically significant abnormal laboratory values for chemistry, hematology and bleeding indices will be graded according to the FDA toxicity scale, or CTCAE if not graded within the FDA scale, and recorded as an AE.
To describe occurrence of adverse events from vital sign measurements following each vaccination. | All study visits (Screening, pre- and post-dose Day 1, Day 8, Day 15, Day 29, pre- and post-dose Day 57, Day64, Day 71, Day 85, pre- and post-dose Day 141, Day 148, Day 156, Day 169, pre- and post-dose Day 225, Day232, Day 253 and Day 337.
  Vital signs assessments will include oral temperature (degrees C) using an oral/tympanic thermometer, respiratory rate (breaths per minute) using manual assessment of breaths, systolic and diastolic blood pressure (mmHg) and heart rate (bpm) using a digital blood pressure machine. Clinically significant abnormal vital sign measurements will be graded according to the FDA toxicity scale, or CTCAE if not graded within the FDA scale, and recorded as an AE.
To determine difference in autologous neutralizing antibody response across dose groups | Pre-vaccinations timepoints (Day 1, Day 57, Day 141 and Day 225), and ~2 weeks after each vaccination (Day15, Day 71, Day 155, and Day 239) and at the EOS (Day 337 post-enrolment).
  Serum will be collected for assessment of occurrence and level of HIV-1-specifi c neutralization titers against vaccine neutralization titers against select Tier 2 panels
To determine difference in heterologous neutralizing antibody response across dose groups | Days 155 and 239. Conditional testing at timepoints (Day 1, Day 57, Day 141 and Day 225), and remaining post-vaccination timepoints (Day 15, Day 71) may be performed
  Serum will be collected for assessment of occurrence and level of HIV-1-specific neutralization titers against select Tier 2 panels

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No